CLINICAL TRIAL: NCT03026673
Title: Hypertension and NSAIDS in the Postpartum Period
Brief Title: Retrospective Review of NSAIDS in the Postpartum Period
Status: Withdrawn | Type: Observational
Why Stopped: staff shortage
Sponsor: St. Louis University (Other)
Responsible Party: Principal Investigator, Jennifer Goldkamp, MD, Principal Investigator, St. Louis University
Other Study IDs: 26975
Record Dates: First submitted 2017-01-18; First posted 2017-01-20 (Estimated); Last update posted 2017-11-13 (Actual); Status verified 2017-11

CONDITIONS: Post Partum Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- NSAID use: The purpose of this study is to establish that NSAIDS are an appropriate analgesic to be used in the postpartum period, and thus women in the immediate postpartum period are the focus of this study.
  Interventions: Other: NSAID use

INTERVENTIONS:
Other: NSAID use — The purpose of the study is to establish that NSAIDS are an appropriate analgesic to be used in the postpartum period, and thus women in the immediate postpartum period are the focus of this study.

SUMMARY:
Chart review of women who have delivered an infant in a single health care system to determine if NSAID use increases blood pressures in the postpartum period.

DETAILED DESCRIPTION:
Nonsteroidal anti-inflammatory drugs (NSAIDs) are the most common medication used for pain relief in the postpartum period in the United States. For pain relief of uterine involution, NSAIDs have shown to be superior to placebo, and equivalent or superior to narcotics. In 2013 the American College of Obstetricians and Gynecologists (ACOG) discouraged the use of NSAIDs in women with pre-eclampsia due to concerns for inadvertently increasing blood pressure. This recommendation is based on non-obstetrics literature, which tended to show a small increase of blood pressures in patients who use NSAIDS. However the literature is mixed, particularly on ibuprofen which is the most common NSAID used in the postpartum. Of the two meta-analysis that are commonly referenced, Pope et al found a decrease of -0.3 (+/- 2.57) mmHg in mean arterial pressure (MAP) in patients with hypertension treated with ibuprofen, and Johnson et al identified an average of 5mmHg increase in blood pressure with ibuprofen use. A large study of 18,325 patients who were treated with NSAIDS or COX-2 inhibitors, found an average of a 2.1 (+/- 0.5) mmHg increase in blood pressure with ibuprofen administration.

There are two articles available in the obstetrics literature on the topic of NSAIDS in women with hypertension disorders. The first is by Makis et al, and is a case series of six women, with discussion of two cases. The explanations of hypertension causes are limited and possible alternate diagnoses are not discussed (6). The second by Wasden et al is a retrospective study of women who had the diagnosis of severe hypertension disorders in pregnancy. The patients were matched 2:1 for women exposed to NSAIDs versus those who did not receive NSAIDs. MAPs were compared, and there was no difference found between the two groups. This second study is better designed and is likely representative of the true outcome of NSAID use in pre-eclamptic women, as the general literature shows a small, non-clinically significant change in blood pressure readings.

ELIGIBILITY:
Inclusion Criteria:

* received NSAIDs post delivery for pain

Exclusion Criteria:

-

Ages: 12 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: pregnant, All ethnic backgrounds will be included.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2017-01-18 (Actual); Primary Completion 2018-04 (Estimated); Study Completion 2019-04 (Estimated)

PRIMARY OUTCOMES:
pain relief | 1 year
  to establish that NSAIDS are an appropriate analgesic to be used in the postpartum period

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Goldkamp, MD, Principal Investigator — St. Louis University
Locations (1):
- St. Mary's Health Center, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No